CLINICAL TRIAL: NCT00339040
Title: Phase II Safety and Immunogenicity Study of Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in HIV Infected Children 7 to 12 Years of Age
Brief Title: Safety of and Immune Response to a Novel Human Papillomavirus Vaccine in HIV Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P1047; 10163 (Registry Identifier: DAIDS ES Registry Number); PACTG P1047
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: HPV
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A: QHPV (Active Comparator): QHPV at week 0, 8, 24, 96.
  Interventions: Biological: Quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like particle (VLP) or Quadrivalent human papillomavirus vaccine (QHPV)
- Arm B: Placebo/QHPV (Other): Placebo at week 0, 8, 24; QHPV at week 96, 104, 120.
  Interventions: Other: Placebo/QHPV

INTERVENTIONS:
Biological: Quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like particle (VLP) or Quadrivalent human papillomavirus vaccine (QHPV) — QHPV at week 0, 8, 24 and 96.
  Other Names: QHPV
  Arms: Arm A: QHPV
Other: Placebo/QHPV — Placebo at week 0, 8, 24 and QHPV at week 96, 104, 120.
  Arms: Arm B: Placebo/QHPV

SUMMARY:
The purpose of this study is to determine the safety of and immune response to a new human papillomavirus (HPV) vaccine in HIV (Human immunodeficiency virus) infected children between the ages of 7 and 12 years.

DETAILED DESCRIPTION:
Genital HPV infection is the most common sexually transmitted infection in the world and may lead to genital warts, anogenital dysplasias, and invasive cancers. HIV infected people and others with compromised immunity are at greater risk for HPV-related complications. In particular, researchers are concerned about the risk of HPV infection to women, who may be infected by their male partners, especially if these partners engage in anal intercourse. HIV infected women tend to have multiple types of HPV (associated with a greater risk of HPV-related disease), are less likely to clear HPV-related conditions, and are more likely to progress to HPV-related disease. The quadrivalent HPV (types 6, 11, 16, 18) L1 virus-like particle (VLP) vaccine to be tested in this study was safe and generally well tolerated in previous studies conducted in healthy and HPV-exposed adolescents, young adults, and older women. However, it is still unclear if the vaccine will be safe and will elicit a similar immune response in younger children. The purpose of this study is to evaluate the safety and immunogenicity of the novel quadrivalent HPV (Types 6, 11, 16, 18) L1 VLP vaccine in HIV infected children 7 to 12 years of age.

This study had two stages and lasted at least 108 weeks. In Stage I, participants were stratified by CD4 percentage (CD4%) nadir and CD4% at study screening (Stratum A: CD4% Nadir < 15 and CD4% ≥ 15 at screening, Stratum B: CD4% Nadir ≥ 15 and < 25 and CD4% ≥ 15 at screening, Stratum C: CD4% Nadir ≥ 25 and CD4% ≥ 25 at screening). Within each stratification group, they were randomly assigned to one of two arms. During Stage I, Arm A (QHPV:Quadrivalent human papillomavirus vaccine) participants received 3 doses of vaccine, while Arm B (Placebo/QHPV) participants received 3 doses of placebo. Participants did not know whether they were receiving vaccine or placebo. Participants received their assigned intervention at study entry and Weeks 8 and 24. At Week 96, Stage II began, and all study participants were told if they received vaccine or placebo in Stage I. Arm A participants received an additional dose of vaccine at Week 96; Arm B participants received doses of vaccine at Weeks 96, 104, and 120. Over the course of the study, there were at least 12 study visits. A physical exam and blood collection occurred at most visits; medical history occurred at selected visits.

After each vaccination, participants were observed for at least 30 minutes to monitor for any allergic reactions possibly resulting from the vaccination. For 15 days following vaccination, parents or guardians were asked to complete a "report card" with details of each child's signs and symptoms. Three days after each vaccination, parents or guardians of study participants were contacted by telephone and asked about any adverse events that a child may have experienced.

ELIGIBILITY:
Inclusion Criteria

Children ages ≥ 7 to < 12 years of age.

A confirmed diagnosis of HIV infection, defined as two positive assays from two different samples. The two results may be in any combination of the following:

* at any age: Deoxyribonucleic acid (DNA) polymerase chain reaction (PCR), Ribonucleic acid (RNA) PCR
* age > 4 weeks: p24 antigen detection
* age >18 months: licensed ELISA (Enzyme-linked immunosorbent assay) with confirmatory Western Blot

CD4% ≥ 15 at the time of screening is required (Note that this is a minimum requirement, and that for Stratum C the CD4% needs to be ≥ 25).

For Strata A and B: Currently stable (≥ 3 months) on highly active antiretroviral therapy (HAART) regimen, defined as three or more antiretrovirals from at least two different therapeutic classes, or therapy with the combination of azidothymidine, lamivudine, and abacavir.

For stratum C no antiretroviral therapy is required.

Parent or legal guardian able and willing to provide signed informed consent.

Negative urine pregnancy test sensitive to 25 International Unit (IU) beta-human chorionic gonadotropin (HCG) for girls who are menstruating (child bearing potential).

Female study volunteers who are participating in sexual activity that could lead to pregnancy must agree to use two reliable methods of contraception, one of which must be a barrier method. A barrier method of contraception (condoms or cervical cap) together with another reliable form of contraception (condoms a , with a spermicidal agent; a diaphragm or cervical cap with spermicide; an intrauterine device [IUD]; or hormonal-based contraception) must be used while on this study. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV-1 transmission

Males participating in the study must not attempt to impregnate a woman, or participate in sperm donation programs. Males engaging in sexual activity that could lead to pregnancy must use a condom.

Exclusion Criteria

Body temperature ≥ 101 F or ≥ 38.3 C, orally determined, within 72 hours prior to the first and each subsequent injection. Subjects may be vaccinated any time in the next seven days thereafter, provided that the site investigator is satisfied that the febrile illness has ended.

Total bilirubin ≥ 5 x Upper Limit of Normal (ULN) at screening.

Alanine transaminase (ALT) or serum glutamic pyruvic transaminase (SGPT) ≥ 5 x ULN at screening in the absence of other explained causes (as determined by the site investigator) at screening.

Serum creatinine ≥ 1.5 mg/dL at screening.

Absolute neutrophil count ≤ 750 cells/mm3 at screening.

Hemoglobin ≤ 9.9 g/dL at screening.

Platelet count ≤ 75,000 cells/mm³ at screening.

Presence of an acute opportunistic non-bacterial or bacterial infection requiring therapy at the time of enrollment; the subject may be entered once he/she is stable on appropriate anti-infective therapy.

Chemotherapy for active malignancy.

Other known or suspected disease of the immune system, or immunosuppressive therapy.

Prior treatment with immunosuppressive or immunomodulation therapy within 60 days of screening.

Prior treatment with three or more week-long courses of corticosteroids (≥ 2.0 mg/kg or ≥ 20 mg total of prednisone-equivalent) within one year of screening; or any systemic (oral or parenteral) steroids (≥ 2.0 mg/kg or ≥ 20 mg total of prednisone-equivalent for ≥ 3 days) within 30 days of study entry.

Prior vaccinations with inactivated vaccines received within two weeks of any dose of study vaccine, and no other vaccinations may be planned for two weeks after each dose of study vaccine.

Prior vaccinations with live vaccines received within three weeks before any dose of study vaccine, and no other vaccinations may be planned for two weeks after each dose of study vaccine.

Prior diagnosis of sexually transmitted infections (STIs), genital warts, or juvenile recurrent papillomatosis.

History of any severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention.

Known allergies to any vaccine component, including aluminum, yeast, or BENZONASE™ (nuclease, Nycomed [used to remove residual nucleic acids from this and other vaccines]).

Previous treatment with any immune globulin preparation or blood-derived products within the six months prior to the first injection and none may be planned during the study.

Known coagulation disorder that would contraindicate Intramuscular (IM) injections.

Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise the outcome of this study.

Breastfeeding.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron J. Levin, MD, Study Chair — Pediatric Infectious Diseases Section, University of Colorado Health Sciences Center
Locations (34):
- United States (32):
  - Usc La Nichd Crs, Alhambra, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. of Orange County, Orange, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Connecticut Children's Med. Ctr., Hartford, Connecticut
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Children's Hosp., New Orleans, Louisiana
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
  - Seattle Children's Hospital CRS, Seattle, Washington
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Ault KA, Giuliano AR, Edwards RP, Tamms G, Kim LL, Smith JF, Jansen KU, Allende M, Taddeo FJ, Skulsky D, Barr E. A phase I study to evaluate a human papillomavirus (HPV) type 18 L1 VLP vaccine. Vaccine. 2004 Aug 13;22(23-24):3004-7. doi: 10.1016/j.vaccine.2004.02.020. PMID 15297048
- [Background] Brown DR, Fife KH, Wheeler CM, Koutsky LA, Lupinacci LM, Railkar R, Suhr G, Barr E, Dicello A, Li W, Smith JF, Tadesse A, Jansen KU. Early assessment of the efficacy of a human papillomavirus type 16 L1 virus-like particle vaccine. Vaccine. 2004 Jul 29;22(21-22):2936-42. doi: 10.1016/j.vaccine.2003.11.059. PMID 15246630
- [Background] Poland GA, Jacobson RM, Koutsky LA, Tamms GM, Railkar R, Smith JF, Bryan JT, Cavanaugh PF Jr, Jansen KU, Barr E. Immunogenicity and reactogenicity of a novel vaccine for human papillomavirus 16: a 2-year randomized controlled clinical trial. Mayo Clin Proc. 2005 May;80(5):601-10. doi: 10.4065/80.5.601. PMID 15887427
- [Result] Levin MJ, Moscicki AB, Song LY, Fenton T, Meyer WA 3rd, Read JS, Handelsman EL, Nowak B, Sattler CA, Saah A, Radley DR, Esser MT, Weinberg A; IMPAACT P1047 Protocol Team. Safety and immunogenicity of a quadrivalent human papillomavirus (types 6, 11, 16, and 18) vaccine in HIV-infected children 7 to 12 years old. J Acquir Immune Defic Syndr. 2010 Oct;55(2):197-204. doi: 10.1097/QAI.0b013e3181de8d26. PMID 20574412
- [Result] P1047 ORAL PRESENTATION at the 25th International Papillomavirus Conference May 8-14 2009, Malmö, Sweden given by Anna Barbara Moscicki. Safety and immunogenicity of Gardasil® in HIV-infected children. Moscicki AB, Weinberg A, Song LY, Handelsman E, Patterson J, Saah A, Radley D, Read JS, Sattler C and Levin MJ for IMPAACT P1047 team.
- [Result] Weinberg A, Song LY, Handelsman E, Moscicki AB, Patterson J, Saah A, Radley D, Esser M, Read J, and Levin MJ for IMPAACT P1047 Team. The P1047 data up to week 28 have been analyzed and presented to 15th CROI as abstract and poster #619a: Safety and Immunogenicity of a Quadrivalent Vaccine to Prevent Human Papilloma Virus (HPV) in HIV-Infected Children: IMPAACT P1047.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 11, 2006 and November 22, 2006 130 participants were enrolled at 34 clinical sites from US & Puerto Rico.
Pre-assignment Details: Participants were stratified by CD4% criteria. Four participants were randomized but did not receive the study treatment. The study analyses were based on 126 participants who received the study treatment.
Groups:
- Arm A QHPV: Participants received three doses of the quadrivalent human papillomavirus vaccine (QHPV) (Types 6, 11, 16, 18) at week 0, 8, and 24 and an additional dose at week 96.
- Arm B Placebo/QHPV: Participants received three doses of the placebo at week 0, 8, and 24 and additional dose of the quadrivalent human papillomavirus vaccine (QHPV) (Types 6, 11, 16, 18) at week 96, 104 and 120.
Period: Stage I
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Started | 96 | 30
Vaccination 1 at Week 0 | 96 | 30
Vaccination 2 at Week 8 | 95 | 30
Vaccination 3 at Week 24 | 94 | 30
Completed | 94 | 29
Not Completed | 2 | 1
Not completed — Not able to attend clinic | 1 | 0
Not completed — Protocol Violation | 1 | 1
Period: Stage II
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Started | 94 | 29
Vaccination 4 at Week 96 | 84 | 29
Vaccination 5 at Week 104 | 0 | 28
Vaccination 6 at Week 120 | 0 | 27
Completed | 84 | 27
Not Completed | 10 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 3 | 0
Not completed — Not able to attend clinic | 1 | 0
Not completed — Site closing | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV | Total
Number analyzed (Participants) | 96 | 30 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (1.4) | 9.9 (1.3) | 9.9 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 18 | 71
  Male | 43 | 12 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 4 | 2 | 6
  Black, non-Hispanic | 54 | 11 | 65
  Hispanic | 37 | 14 | 51
  Others | 1 | 3 | 4
Stratification groups [Number; unit: participants] — STRATIFICATION: Participant were stratified by CD4% criteria into three strata:
  * Stratum A: CD4% Nadir < 15 and CD4% ≥ 15 at screening
  * Stratum B: CD4% Nadir ≥ 15 and < 25 and CD4% ≥ 15 at screening
  * Stratum C: CD4% Nadir ≥ 25 and CD4% ≥ 25 at screening
  participants
    Stratum A | 31 | 10 | 41
    Stratum B | 32 | 11 | 43
    Stratum C | 33 | 9 | 42
CD4 count [Mean (Standard Deviation); unit: cells/µL] | 868 (367) | 1013 (455) | 903 (393)
CD4% [Mean (Standard Deviation); unit: percentage of total lymphocytes] | 33.9 (7.9) | 35.8 (8.6) | 34.3 (8.1)
Log10(RNA) [Mean (Standard Deviation); unit: Log10(copies/mL)] | 2.7 (0.9) | 2.6 (0.8) | 2.7 (0.9)
RNA group [Number; unit: participants]
  ≤400 copies/mL | 65 | 22 | 87
  401 to ≤5000 copies/mL | 16 | 5 | 21
  >5000 copies/mL | 15 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Developing Grade 3 or 4 Adverse Events (AEs)
Description: Adverse events were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (December 2004). The grades used are: Grade 1="Mild", Grade 2="Moderate", Grade 3="Severe", Grade 4="Potentially Life-Threatening". All grade 3 and higher signs, symptoms, and laboratory toxicities were included.
Time Frame: Within 14 days of first three doses of vaccination
Population: Any participant who received at least one study vaccine/placebo were included in the safety analysis.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Number analyzed (Participants) | 96 | 30
percent of participants | 7.3 [3.0 to 14.5] | 6.7 [0.8 to 22.1]
Statistical Analysis 1: Comparison: Arm A QHPV vs Arm B Placebo/QHPV; Test type: Superiority or Other; p = 1.00, Fisher Exact

2. Primary Outcome: Percent of Participants Developing Grade 3 or 4 Adverse Events (AEs) Attributed to Study Treatment
Description: Adverse events were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (December 2004). All grade 3 and higher signs, symptoms, and laboratory toxicities attributed to study treatment were included. The relationship between the Adverse Events and the vaccination were evaluated by study team and assigned to, for example, "Treatment related", "Non-treatment related", "Baseline", "Possibly treatment related".
Time Frame: Within 14 days of first three doses of vaccination
Population: Any participant who received at least one study vaccine/placebo were included in the safety analysis
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Number analyzed (Participants) | 96 | 30
percent of participants | 0 [0 to 0] | 0 [0 to 0]

3. Primary Outcome: Percent of Participants With Human Papillomavirus (HPV) Type-Specific Seroconversion
Description: Serum anti-HPV 6, 11, 16, and 18 antibody was measured using a competitive Luminex immunoassay (cLIA; reported in milli-Merck Units [mMU]/mL). Sero-positivity was defined as an anti-HPV titer ≥20, 16, 20, and 24 mMU/mL, for HPV types 6, 11, 16, and 18, respectively.
Time Frame: At week 28 after beginning the vaccination series
Population: The type-specific results are reported for participants remaining after exclusion of those with protocol violations, unevaluable specimens, or the presence of type-specific sero-positive antibody at baseline.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Number analyzed (Participants) | 96 | 30
percent of participants
  Serotype 6: number analyzed (Participants) | 87 | 27
  Serotype 6 | 100.0 [95.9 to 100.0] | 0.0 [0.0 to 12.8]
  Serotype 11: number analyzed (Participants) | 90 | 27
  Serotype 11 | 100.0 [95.9 to 100.0] | 0.0 [0.0 to 12.8]
  Serotype 16: number analyzed (Participants) | 90 | 27
  Serotype 16 | 100.0 [95.9 to 100.0] | 3.7 [0.1 to 19.0]
  Serotype 18: number analyzed (Participants) | 90 | 27
  Serotype 18 | 96.7 [90.6 to 99.3] | 0.0 [0.0 to 12.8]

4. Primary Outcome: Serum Anti-HPV Antibody Titers (cLIA)
Description: Geometric means of Type-specific Serum anti-HPV antibody titers (cLIA)
Time Frame: Arm A week 0, 28, 72, 96, 97, 100; Arm B week 0, 28, 72, 96, 97, 100, 124.
Population: The type-specific results are reported for participants remaining after exclusion of those with protocol violations, unevaluable specimens, or the presence of type-specific sero-positive antibody at baseline as well as any participants with any missing values at any time points.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-Merck units [mMU]/mL
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Number analyzed (Participants) | 96 | 30
milli-Merck units [mMU]/mL
  Serotype 6 study entry: number analyzed (Participants) | 69 | 23
  Serotype 6 study entry | 3.8 [3.5 to 4.1] | 4.1 [3.4 to 4.9]
  Serotype 6 week 28: number analyzed (Participants) | 69 | 23
  Serotype 6 week 28 | 544.2 [395.4 to 749.1] | 4.5 [3.7 to 5.4]
  Serotype 6 week 72: number analyzed (Participants) | 69 | 23
  Serotype 6 week 72 | 256.4 [196.5 to 334.7] | 4.3 [3.6 to 5.1]
  Serotype 6 week 96: number analyzed (Participants) | 69 | 23
  Serotype 6 week 96 | 227.9 [167.3 to 310.3] | 4.5 [3.6 to 5.8]
  Serotype 6 week 97: number analyzed (Participants) | 69 | 23
  Serotype 6 week 97 | 1604.8 [1162.0 to 2216.1] | 17.1 [7.1 to 41.5]
  Serotype 6 week 100: number analyzed (Participants) | 69 | 23
  Serotype 6 week 100 | 2473.6 [1770.2 to 3456.4] | 79.7 [43.7 to 145.3]
  Serotype 6 week 124: number analyzed (Participants) | 0 | 23
  Serotype 6 week 124 |  | 678.8 [396.4 to 1162.2]
  Serotype 11 study entry: number analyzed (Participants) | 72 | 23
  Serotype 11 study entry | 4.1 [3.9 to 4.2] | 4.0 [4.0 to 4.0]
  Serotype 11 week 28: number analyzed (Participants) | 72 | 23
  Serotype 11 week 28 | 1396.6 [1103.8 to 1767.1] | 4.2 [3.8 to 4.7]
  Serotype 11 week 72: number analyzed (Participants) | 72 | 23
  Serotype 11 week 72 | 313.1 [234.4 to 418.3] | 4.1 [3.9 to 4.5]
  Serotype 11 week 96: number analyzed (Participants) | 72 | 23
  Serotype 11 week 96 | 286.5 [207.1 to 396.4] | 4.0 [4.0 to 4.0]
  Serotype 11 week 97: number analyzed (Participants) | 72 | 23
  Serotype 11 week 97 | 1931.7 [1389.1 to 2686.3] | 11.8 [5.5 to 25.6]
  Serotype 11 week 100: number analyzed (Participants) | 72 | 23
  Serotype 11 week 100 | 3611.2 [2746.8 to 4747.6] | 86.4 [48.7 to 153.6]
  Serotype 11 week 124: number analyzed (Participants) | 0 | 23
  Serotype 11 week 124 |  | 1023.0 [704.2 to 1486.0]
  Serotype 16 study entry: number analyzed (Participants) | 71 | 23
  Serotype 16 study entry | 5.5 [5.5 to 5.5] | 5.5 [5.5 to 5.5]
  Serotype 16 week 28: number analyzed (Participants) | 71 | 23
  Serotype 16 week 28 | 5172.5 [3889.8 to 6878.2] | 5.7 [5.3 to 6.2]
  Serotype 16 week 72: number analyzed (Participants) | 71 | 23
  Serotype 16 week 72 | 1126.4 [788.6 to 1609.0] | 5.5 [5.5 to 5.5]
  Serotype 16 week 96: number analyzed (Participants) | 71 | 23
  Serotype 16 week 96 | 1034.5 [708.8 to 1509.7] | 5.5 [5.5 to 5.5]
  Serotype 16 week 97: number analyzed (Participants) | 71 | 23
  Serotype 16 week 97 | 6167.8 [4391.8 to 8661.8] | 12.1 [5.4 to 27.1]
  Serotype 16 week 100: number analyzed (Participants) | 71 | 23
  Serotype 16 week 100 | 11205.6 [8184.7 to 15341.5] | 142.6 [74.1 to 274.5]
  Serotype 16 week 124: number analyzed (Participants) | 0 | 23
  Serotype 16 week 124 |  | 4113.8 [2404.2 to 7039.3]
  Serotype 18 study entry: number analyzed (Participants) | 71 | 23
  Serotype 18 study entry | 5.1 [4.9 to 5.3] | 5.0 [5.0 to 5.0]
  Serotype 18 week 28: number analyzed (Participants) | 71 | 23
  Serotype 18 week 28 | 931.2 [616.7 to 1406.0] | 5.0 [5.0 to 5.0]
  Serotype 18 week 72: number analyzed (Participants) | 71 | 23
  Serotype 18 week 72 | 148.2 [92.5 to 237.4] | 5.0 [5.0 to 5.0]
  Serotype 18 week 96: number analyzed (Participants) | 71 | 23
  Serotype 18 week 96 | 142.0 [86.6 to 232.8] | 5.0 [5.0 to 5.0]
  Serotype 18 week 97: number analyzed (Participants) | 71 | 23
  Serotype 18 week 97 | 925.7 [567.6 to 1510.0] | 7.1 [4.6 to 11.0]
  Serotype 18 week 100: number analyzed (Participants) | 71 | 23
  Serotype 18 week 100 | 1530.7 [991.7 to 2362.4] | 18.7 [10.6 to 32.8]
  Serotype 18 week 124: number analyzed (Participants) | 0 | 23
  Serotype 18 week 124 |  | 734.3 [357.3 to 1508.8]

5. Secondary Outcome: CD4 Count Over Time
Time Frame: Arm A week 0, 8, 12, 24, 28, 72, 96, 100 and 108; Arm B week 0, 8, 12, 24, 28, 72, 96, 100, 104, 108, 120, and 124.
Population: Any participant who received at least one study vaccine/placebo and with non-missing CD4 counts at the respective time point.
Measure: Mean (95% Confidence Interval); unit: cells/µL
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Number analyzed (Participants) | 96 | 30
cells/µL
  CD4 count at study entry | 868 [794 to 942] | 1013 [843 to 1183]
  CD4 count at week 8: number analyzed (Participants) | 93 | 30
  CD4 count at week 8 | 907 [830 to 985] | 1018 [851 to 1185]
  CD4 count at week 12: number analyzed (Participants) | 93 | 30
  CD4 count at week 12 | 906 [828 to 983] | 1056 [830 to 1282]
  CD4 count at week 24: number analyzed (Participants) | 94 | 30
  CD4 count at week 24 | 864 [792 to 936] | 993 [826 to 1160]
  CD4 count at week 28: number analyzed (Participants) | 95 | 30
  CD4 count at week 28 | 875 [800 to 950] | 959 [803 to 1115]
  CD4 count at week 72: number analyzed (Participants) | 88 | 30
  CD4 count at week 72 | 823 [746 to 900] | 933 [768 to 1098]
  CD4 count at week 96: number analyzed (Participants) | 88 | 30
  CD4 count at week 96 | 781 [712 to 849] | 874 [718 to 1031]
  CD4 count at week 100: number analyzed (Participants) | 85 | 29
  CD4 count at week 100 | 831 [754 to 907] | 924 [766 to 1083]
  CD4 count at week 104: number analyzed (Participants) | 0 | 27
  CD4 count at week 104 |  | 929 [776 to 1082]
  CD4 count at week 108: number analyzed (Participants) | 82 | 28
  CD4 count at week 108 | 839 [757 to 921] | 980 [786 to 1174]
  CD4 count at week 120: number analyzed (Participants) | 0 | 28
  CD4 count at week 120 |  | 931 [745 to 1117]
  CD4 count at week 124: number analyzed (Participants) | 0 | 27
  CD4 count at week 124 |  | 920 [728 to 1112]

6. Secondary Outcome: CD4 Percent Over Time
Time Frame: Arm A week 0, 8, 12, 24, 28, 72, 96, 100 and 108; Arm B week 0, 8, 12, 24, 28, 72, 96, 100, 104, 108, 120, and 124.
Population: Any participant who received at least one study vaccine/placebo and with non-missing CD4%.
Measure: Mean (95% Confidence Interval); unit: percentage of total lymphocytes
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Number analyzed (Participants) | 96 | 30
percentage of total lymphocytes
  CD4 percent at study entry | 34 [32 to 35] | 36 [33 to 39]
  CD4 percent at week 8: number analyzed (Participants) | 93 | 30
  CD4 percent at week 8 | 34 [32 to 35] | 36 [33 to 39]
  CD4 percent at week 12: number analyzed (Participants) | 93 | 30
  CD4 percent at week 12 | 35 [33 to 37] | 37 [33 to 41]
  CD4 percent at week 24: number analyzed (Participants) | 94 | 30
  CD4 percent at week 24 | 34 [33 to 36] | 35 [31 to 39]
  CD4 percent at week 28: number analyzed (Participants) | 95 | 30
  CD4 percent at week 28 | 34 [33 to 36] | 34 [31 to 38]
  CD4 percent at week 72: number analyzed (Participants) | 88 | 30
  CD4 percent at week 72 | 33 [32 to 35] | 34 [30 to 38]
  CD4 percent at week 96: number analyzed (Participants) | 88 | 30
  CD4 percent at week 96 | 33 [32 to 35] | 34 [30 to 38]
  CD4 percent at week 100: number analyzed (Participants) | 85 | 29
  CD4 percent at week 100 | 35 [33 to 37] | 35 [32 to 39]
  CD4 percent at week 104: number analyzed (Participants) | 0 | 27
  CD4 percent at week 104 |  | 36 [32 to 40]
  CD4 percent at week 108: number analyzed (Participants) | 82 | 28
  CD4 percent at week 108 | 35 [33 to 37] | 34 [30 to 38]
  CD4 percent at week 120: number analyzed (Participants) | 0 | 28
  CD4 percent at week 120 |  | 37 [32 to 42]
  CD4 percent at week 124: number analyzed (Participants) | 0 | 27
  CD4 percent at week 124 |  | 35 [31 to 39]

7. Secondary Outcome: HIV-1 Viral Load (Ribonucleic Acid [RNA] Copies/ml) Over Time
Time Frame: Arm A week 0, 8, 12, 24, 28, 72, 96, 100 and 108; Arm B week 0, 8, 12, 24, 28, 72, 96, 100, 104, 108, 120, and 124.
Population: Any participant who received at least one study vaccine/placebo and with non-missing HIV-1 viral load at the respective time point.
Measure: Log Mean (95% Confidence Interval); unit: Log10 (copies/mL)
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Number analyzed (Participants) | 96 | 30
Log10 (copies/mL)
  Log10(RNA) at study entry | 2.7 [2.5 to 2.9] | 2.6 [2.3 to 2.9]
  Log10(RNA) at week 8: number analyzed (Participants) | 92 | 30
  Log10(RNA) at week 8 | 2.8 [2.6 to 3.0] | 2.8 [2.5 to 3.1]
  Log10(RNA) at week 12: number analyzed (Participants) | 93 | 30
  Log10(RNA) at week 12 | 2.7 [2.6 to 2.9] | 2.8 [2.5 to 3.2]
  Log10(RNA) at week 24: number analyzed (Participants) | 94 | 29
  Log10(RNA) at week 24 | 2.8 [2.6 to 2.9] | 2.7 [2.4 to 3.1]
  Log10(RNA) at week 28: number analyzed (Participants) | 95 | 30
  Log10(RNA) at week 28 | 2.7 [2.6 to 2.9] | 2.8 [2.4 to 3.1]
  Log10(RNA) at week 72: number analyzed (Participants) | 87 | 30
  Log10(RNA) at week 72 | 2.7 [2.5 to 2.8] | 2.7 [2.4 to 3.1]
  Log10(RNA) at week 96: number analyzed (Participants) | 88 | 28
  Log10(RNA) at week 96 | 2.6 [2.4 to 2.8] | 2.4 [2.1 to 2.6]
  Log10(RNA) at week 100: number analyzed (Participants) | 84 | 29
  Log10(RNA) at week 100 | 2.6 [2.4 to 2.8] | 2.4 [2.1 to 2.6]
  Log10(RNA) at week 104: number analyzed (Participants) | 0 | 27
  Log10(RNA) at week 104 |  | 2.4 [2.0 to 2.7]
  Log10(RNA) at week 108: number analyzed (Participants) | 87 | 28
  Log10(RNA) at week 108 | 2.6 [2.4 to 2.7] | 2.5 [2.1 to 2.8]
  Log10(RNA) at week 120: number analyzed (Participants) | 0 | 28
  Log10(RNA) at week 120 |  | 2.3 [2.0 to 2.6]
  Log10(RNA) at week 124: number analyzed (Participants) | 0 | 27
  Log10(RNA) at week 124 |  | 2.3 [1.9 to 2.6]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time when participants started to receive study treatment until study completion and before August 10, 2009 (primary completion date).
Description: Expedited adverse event (AE) reporting followed Intensive Division of AIDS (DAIDS) Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities, requiring hospitalization, and >=grade 3 AEs defined by the "DAIDS Table for Grading the Severity of Adult and Pediatric AEs", V1.0, 12/2004.
Arm/Group | Arm A QHPV | Arm B Placebo/QHPV
Serious Adverse Events (participants affected / at risk) | 5/96 | 2/30
Other Adverse Events (participants affected / at risk) | 93/96 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A QHPV (N=96) | Arm B Placebo/QHPV (N=30)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 1
Blood amylase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A QHPV (N=96) | Arm B Placebo/QHPV (N=30)
Ear pain (Ear and labyrinth disorders) | 5 | 3
Conjunctivitis (Eye disorders) | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 9 | 4
Chest pain (General disorders) | 5 | 0
Gait disturbance (General disorders) | 0 | 2
Injection site pain (General disorders) | 13 | 2
Pyrexia (General disorders) | 14 | 10
Acute sinusitis (Infections and infestations) | 4 | 5
Gastroenteritis (Infections and infestations) | 7 | 0
Otitis media acute (Infections and infestations) | 4 | 3
Pharyngitis (Infections and infestations) | 5 | 3
Pharyngitis streptococcal (Infections and infestations) | 3 | 3
Pneumonia (Infections and infestations) | 2 | 2
Purulent discharge (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 20 | 6
Aspartate aminotransferase increased (Investigations) | 15 | 10
Blood albumin abnormal (Investigations) | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 14 | 1
Blood bicarbonate abnormal (Investigations) | 21 | 5
Blood bilirubin increased (Investigations) | 11 | 6
Blood cholesterol increased (Investigations) | 17 | 4
Blood creatinine increased (Investigations) | 5 | 3
Blood glucose decreased (Investigations) | 37 | 10
Blood glucose increased (Investigations) | 12 | 7
Blood phosphorus decreased (Investigations) | 7 | 1
Blood potassium decreased (Investigations) | 12 | 3
Blood sodium decreased (Investigations) | 28 | 11
Blood triglycerides increased (Investigations) | 7 | 0
Haemoglobin decreased (Investigations) | 5 | 1
Neutrophil count decreased (Investigations) | 36 | 10
Platelet count decreased (Investigations) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 6 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and Merck & Co., Inc., NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.